CLINICAL TRIAL: NCT07297225
Title: Metabolic Dysfunction-Associated Fatty Liver Disease Impairs Intraoperative Indocyanine Green Fluorescence Cholangiography Quality: Development and Validation of a Predictive Model
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-KY-323
Record Dates: First submitted 2025-09-21; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: MAFLD; Cholecystitis; Gallbladder Polyps; Cholelithiasis
MeSH Terms: conditions — Cholecystitis; Cholelithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Non-MAFLD Group
  Interventions: Other: Retrospective observational study without intervention measures
- MAFLD Group
  Interventions: Other: Retrospective observational study without intervention measures
- Training Cohort
  Interventions: Other: Retrospective observational study without intervention measures
- Validation Cohort
  Interventions: Other: Retrospective observational study without intervention measures

INTERVENTIONS:
Other: Retrospective observational study without intervention measures — Retrospective observational study without intervention measures

SUMMARY:
Near-infrared fluorescence cholangiography has been shown to improve the clinical outcomes of laparoscopic cholecystectomy (LC). However, it remains unclear whether hepatic steatosis in patients with metabolic dysfunction-associated fatty liver disease (MAFLD) influences the quality of indocyanine green fluorescence imaging (ICG-FI), and whether the quality can be predicted preoperatively. This study aimed to evaluate the impact of MAFLD on intraoperative fluorescence quality and to develop a multiple linear regression model for predicting intraoperative ICG-FI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, any sex;
2. Definite surgical indication for cholecystectomy;
3. Underwent LC;
4. No severe contraindications such as significant cardiac, pulmonary, renal, or cerebral dysfunction.

Exclusion Criteria:

1. Known allergy to ICG or iodinated contrast agents;
2. Use of medications affecting biliary excretion within 2 weeks prior to surgery; (3) LC without ICG-FI;

(4) Incomplete clinical data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) Age 18-75 years, any sex; (2) Definite surgical indication for cholecystectomy; (3) Underwent LC; (4) No severe contraindications such as significant cardiac, pulmonary, renal, or cerebral dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Common bile duct FI / Liver background FI (C/L) | Perioperative period
  The common bile duct-to-liver background fluorescence intensity ratio (C/L) [Unit: Dimensionless number] [Time Frame: Perioperative period] [Measurement steps: Three photographs per case were obtained with the following requirements: Calot's triangle centred in the image, liver background positioned superiorly, and the CBD inferiorly, ensuring all measurement sites were visible and unobstructed. Each image was converted to greyscale, and regions of interest (ROI) of >3000 pixels were selected for each critical structure to calculate FI. The mean FI from the three images was recorded as the final value for each structure.]

SECONDARY OUTCOMES:
Qualitative assessment of fluorescence visualization | Perioperative period
  Qualitative assessment of fluorescence visualization. [Time Frame: Perioperative period] [Unit: Dimensionless number] [Measurement steps: It was performed by three senior surgeonsScores were averaged and graded on a five-point scale adapted from previous studies (1=completely invisible, impairs visualization; 2=poor, faint fluorescence, no added value; 3= visible but blurred, some added value; 4=good, clear visualization with significant added value; 5= excellent, very clear visualization with typical added value)]

OTHER OUTCOMES:
Preoperative laboratory test indicators and baseline data | Perioperative period
  HSI（Hepatic Steatosis Index) and FSI (Framingham Steatosis Index) [Time Frame: Perioperative period] [Unit: Dimensionless number] [The variables included：ALT and AST(IU/L), BMI(kg/m2), gender(male/female), diabete(yes/no), age(years), TG (mmol/L), Hypertension(yes/no)]

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China